CLINICAL TRIAL: NCT02158832
Title: Rehabilitation of Breast Cancer Treatment Related Lymphedema Using Electro-acupuncture: A Randomized Controlled Trial
Brief Title: Acupuncture for Lymphedema Secondary to Breast Cancer Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study Principal Investigator relocated and the grant funding the trial expired.
Sponsor: McMaster University (Other)
Collaborators: Canadian Interdisciplinary Network Complementary & Alternative Medicine Research (Other); Holistic Health Research Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIREB 14-089
Record Dates: First submitted 2014-05-14; First posted 2014-06-09 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Lymphedema
Keywords: Lymphoedema; Edema; Oedema; Cancer; Breast Cancer
MeSH Terms: conditions — Lymphedema; Edema; Neoplasms; Breast Neoplasms | interventions — Acupuncture Therapy; Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture + Electrical Stimulation (Experimental): Acupuncture needles are inserted beneath the skin and electrical stimulation applied for 20 minutes.
  Interventions: Device: Acupuncture + Electrical Stimulation
- Control (No Intervention): Participants who are randomized to receive no intervention will still receive physical assessment.

INTERVENTIONS:
Device: Acupuncture + Electrical Stimulation — 2 acupuncture needles are inserted into the upper back. 10Hz, 0.5ms biphasic square wave electrical pulses are applied to needles x20 mins. Current >sensation threshold & maintained at a level that is comfortable/painless & does not elicit skeletal muscle contractions (~5mA, <10mA).
  Needle locations are in the vicinity of nerves that supply the affected upper limb:
  EX-B1': Affected hemisphere, 1.5cm lateral to C5 spinous process. Insertion angle: shallow, 'inferior-lateral', ~15⁰ perpendicular to the skin, ~15⁰ lateral to the midline. Depth: ~1.5 cm (secure anchorage).
  EX-HN15': Affected hemisphere, 1.5cm lateral to the C7 spinous process. Insertion angle: shallow, 'inferior-medial' ~15⁰ perpendicular to the skin, ~15⁰ medial. Depth: ~1.5 cm (secure anchorage).
  Other Names: Acupuncture; Electrical Stimulation; Electro-Acupuncture
  Arms: Acupuncture + Electrical Stimulation

SUMMARY:
This study is being conducted to determine if electro-acupuncture can reduce swelling of the arm due to breast cancer treatment (commonly referred to as 'lymphedema'). Research conducted on animals suggests that such treatment might be used to improve circulation leading to reductions in swelling. Previous research in humans with lymphedema suggests that treatment may be safe to use, although results regarding its efficacy in the reduction of swelling have not yet been established.

This research will use sophisticated, non-invasive assessment methods to determine if a single session of electro-acupuncture treatment can be effective for reducing lymphedema. Results may be used to further develop our understanding of how electro-acupuncture can be used in the management of this condition. Electro-acupuncture may provide a promising complement or alternative to conventional lymphedema treatments such as compression bandaging, massage therapy or surgery.

DETAILED DESCRIPTION:
Participants will be invited to attend a 30-60 minute screening visit to determine eligibility. This screening visit will be located at a laboratory at McMaster University's Institute of Applied Health Sciences. Eligibility will be determined using health questionnaires and non-invasive physical assessment of the upper limbs. Participants may not be eligible for further participation based on their health status and risks to health and safety.

Participants meeting eligibility criteria will be invited to 1 scheduled appointment (30-60 minutes in duration). The appointment time will be scheduled according to individual symptoms, such that it will coincide with the time of day that lymphedema symptoms are predicted to be at their highest. Upon arrival at the scheduled appointment, participants will be randomized to receive 20 minutes of acupuncture+applied electrical stimulation or no treatment. Participants in both groups will be asked to provide physical assessment data over a period of 30 minutes during the scheduled appointment. Differences between groups in tissue swelling of the affected upper-limb will be determined immediately following treatment, and at 10 minutes following treatment.

Participants will be asked to report any significant changes to their health state for a period of 2 weeks following treatment. A follow-up questionnaire will be made available at 2 weeks following attendance of the scheduled appointment.

ELIGIBILITY:
Inclusion Criteria:

* >1yr following the conclusion of breast cancer treatment
* Lymphedema of the upper limb: unilateral (one-side)

Exclusion Criteria:

* History or evidence of hormone-receptor positive cancer
* Previous nodal dissection or radiotherapy to other regions
* Contraindications for acupuncture or electrical stimulation
* Pre-cancer or bi-lateral lymphedema
* Evidence of active cancer
* History of contralateral cancer, radiation or surgery
* Edema of the neck/midline/torso
* Pregnancy
* Allergies to nickel, chromium, or silicon
* Seizures (epilepsy)
* Tremors (shakiness) that may interfere with treatment
* Infections, scarring, open wounds, or broken skin at needle sites
* Infections, open wounds, or broken skin on the upper limbs (electrode & landmark sites)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04 (Estimated); Primary Completion 2017-01 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in amount of arm tissue water determined by Bioimpedance Analysis | Before and after a 20 minute period at a single scheduled appointment
  Bioimpedance analysis devices take readings using 8 electrode pads that are placed on top of the skin of the arms. The electrode pads are connected to a computer that transmits a small amount of electrical current between the electrode pads. The process of taking readings takes less than 1 minute and is painless (participants may not be able to feel it working).

SECONDARY OUTCOMES:
Change in dermal concentration of red blood cells in the arm assessed using light polarization spectroscopy | Repeated measures during a single scheduled appointment - once every 2 minutes for 44 minutes
  A digital camera is used to 'see under the skin' and measure the amount of red blood cells in the arm. The camera is an ordinary digital camera connected to special computer software. Assessment using the camera is harmless and patients will not be able to feel it working. A series of digital photographs of a small area of the arms will be taken. The computer uses these photographs to calculate a number that represents the amount of blood contained in the skin of the arm.
Change in arm circumference | Before and after a 20 minute period at a single scheduled appointment
  Measurements are taken of both arms using a flexible measuring tape to be used in the calculation of size and volume.
Lymphedema Questionnaire | Administered at a single screening visit and 2 week follow up
  Survey is administered to collect data pertaining to the condition of lymphedema.

OTHER OUTCOMES:
Baseline current perception threshold | Readings are taken once during a 15 minute during a single screening visit
  Small electrodes will be placed on the tips of the middle finger and a weak electrical stimulus applied. This electrical stimulus will be raised up until the point participants can feel it as a 'tingling' or 'tapping' sensation (a non-painful stimulus). Doing so is used to assess the functioning of nerves in the affected arm.
Baseline arm tissue water determined by Bioimpedance Analysis | Readings are taken once during a 15 minute screening visit
  Bioimpedance analysis devices take readings using 8 electrode pads that are placed on top of the skin of the arms. The electrode pads are connected to a computer that transmits a small amount of electrical current between the electrode pads. The process of taking readings takes less than 1 minute and is painless (participants may not be able to feel it working).

CONTACTS AND LOCATIONS:
Overall Officials: Derek Rosa, PhD(c), Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada